CLINICAL TRIAL: NCT07074782
Title: Retinal Ganglion Cell Neuroprotection Under Prostaglandin Analogues: NEUROPA - a Retrospective Cohort Study
Brief Title: Retinal Ganglion Cell Neuroprotection Under Prostaglandin Analogues
Acronym: NEUROPA
Status: Not yet recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-GLC-2025-18
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group (Non-Prostaglandin IOP-lowering compound): 750 eyes treated with intraocular pressure-lowering compounds that do not belong to the prostaglandin analogue class. These treatments may include beta-adrenergic blocking agents (e.g., timolol, betaxolol), carbonic anhydrase inhibitors (e.g., dorzolamide, brinzolamide), alpha-2 adrenergic agonists (e.g., brimonidine) or rho kinase inhibitors (e.g., netarsudil).
- Interventional group (prostaglandin analogues): 750 eyes treated with any prostaglandin analogue, such as latanoprost (e.g., Xalatan® 50 µg/mL, Pfizer), travoprost, tafluprost, bimatoprost, or unoprostone.

SUMMARY:
The goal of this observational study is to evaluate whether prostaglandin analogue eye drops have a direct neuroprotective effect on retinal ganglion cells - beyond their intraocular pressure (IOP)-lowering effect - in adult patients with glaucoma or ocular hypertension. The study includes individuals diagnosed with glaucoma (any sex/gender, adult age groups) undergoing standard clinical treatment. The main questions it aims to answer are:

* Do prostaglandin analogues provide a neuroprotective effect on retinal ganglion cells that is independent of their IOP-lowering properties?
* Should prostaglandin analogues be promoted/favoured over other IOP-lowering compounds for long-term glaucoma management?

Researchers will compare an interventional group, which consist of 750 eyes treated with prostaglandin analogues (e.g., latanoprost, travoprost, tafluprost, bimatoprost, unoprostone), with a control group, which consist of 750 eyes treated with non-prostaglandin IOP-lowering compounds (e.g., timolol, dorzolamide, brimonidine, netarsudil) to see if treatment with prostaglandin analogues is associated with better retinal ganglion cell survival over a period of 3 years (36 months).

Data will be collected from individuals who had at least 36 months of documented follow-up, with clinical data available at approximately 3, 6, 12, 24, and 36 months. Eligible individuals must have been treated with either prostaglandin analogues or other intraocular pressure (IOP)-lowering agents as part of routine clinical care. The data to be obtained from medical records will include at least:

* Intraocular pressure readings
* Visual field testing
* OCT measures
* Visual acuity
* Adverse events
* Treatment adherence/compliance
* Additional glaucoma interventions

DETAILED DESCRIPTION:
Glaucoma is among the most prevalent causes of irreversible blindness and is characterized by a progressive, irreversible degeneration of the retinal ganglion cells. Elevated intraocular pressure (IOP) is the most important glaucoma risk factor and the only risk factor that is readily modifiable with established treatment options, which include pharmacological approaches, laser treatment, and surgery. However, in many patients the disease progresses even after IOP is effectively lowered. Hence, neuroprotective treatment approaches that go beyond IOP lowering are needed.

Prostaglandin analogue eye drops reduce IOP by increasing uveoscleral outflow and are a well-established treatment option in ocular hypertension and glaucoma. Animal studies suggest that prostaglandin analogues may have a direct neuroprotective effect on retinal ganglion cells in addition to the effect mediated by IOP lowering. Proposed mechanisms of action include inhibiting of caspase-3 and cyclooxygenase as well as activation of polypeptide 2B1 and Klotho protein. However, this proposed additional, direct neuroprotective effect has not yet been tested in human patients. The viability and functional status of the retinal ganglion cells in glaucoma can be assessed by morphological readings, the standard nowadays being various optical coherence tomography modalities, and by visual field testing. Detection of Apoptosing Retinal Cells (DARC) is another, relatively novel technology that allows for quantification of retinal ganglion cell death, presumably on a much shorter time scale.

This is an observational, retrospective and longitudinal clinical study, according to the normal clinical practice.

This study aims to evaluate prostaglandin analogues neuroprotective effect on retinal ganglion cells apart from intraocular pressure (IOP)-lowering over a period of 3 years (36 months) and whether treatment of ocular hypertension and glaucoma participants with prostaglandin analogues should be promoted/ favoured over other IOP-lowering compounds. It will have a follow-up at 3, 6, 12, 24, and 36 months in eyes with glaucoma treated with prostaglandin analogues or a different topically applied compound.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Established glaucoma diagnosis (primary open-angle glaucoma, normal tension Glaucoma, pseudoexfoliation glaucoma, pigmentary dispersion glaucoma) in either eye
* Visual field mean deviation (MD; location-weighted mean difference from average age-corrected visual field sensitivity) of 2 visual fields differing by no more than 3 dB, for a mean deviation of better than -6.0 dB, or by no more than 4 dB, for a mean deviation worse than -6.0 dB, as measured using Humphrey perimetry (or equivalent Haag-Streit / Octopus; in at least one eye; analogous to The United Kingdom Glaucoma Treatment Study)
* Treatment with either prostaglandin analogues only or another topically applied IOP-lowering compound only for at least 3 years
* Documented follow-up period of at least 3 years
* At least 6 patient visits documented over the follow-up period with readings of IOP, visual field, OCT
* No additional glaucoma intervention apart from laser trabeculoplasty and/or cataract surgery during the observational period

Exclusion Criteria:

* Follow-up period < 3 years
* Number of patient visits <6 visits
* Number of OCT, visual field readings during the observation period < 6
* Low compliance/therapy interruption
* Beginning of combination therapy of prostaglandin analogues and other IOP lowering eye drops during the observation period
* In case of glaucoma diagnosis in both eyes: different topical IOP-lowering treatment regimes (e.g. prostaglandin analogues in one eye and beta-adrenergic blocking agents in the fellow eye)
* Additional glaucoma intervention during the observational period other than laser trabeculoplasty and/or cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1500 eyes (750 treated with prostaglandin analogues and 750 treated with a different IOP-lowering compound)
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP), measured using a Goldmann applanation tonometer, an iCare tonometer, or similar. Change in IOP value (mmHg). | 6 months
  Change in IOP value (mmHg).
Visual field (VF) - Mean Deviation, measured by automated perimetry testing devices, such as Haag-Streit Octopus, Zeiss Humphrey, or similar | 6 months
  Evaluation of Change in Mean Deviation (MD, dB).
Visual Field - Pattern Standard Deviation, measured by automated perimetry testing devices, such as Haag-Streit Octopus, Zeiss Humphrey, or similar. | 6 months
  Evaluation of Pattern Standard Deviation (PSD, dB).
Visual Field - Glaucoma Progression Analysis (GPA), measured by automated perimetry testing devices, such as Haag-Streit Octopus, Zeiss Humphrey, or similar. | 6 months
  Evaluation of Glaucoma Progression Analysis (GPA, %/year).
Optical Coherence Tomography - Change in Average GCL+IPL Thickness, measured by Heidelberg Spectralis, Zeiss Cirrus, or similar. | 6 months
  Evaluation of Change in Average GCL+IPL thickness (µm).
Optical Coherence Tomography - Average RNFL Thickness, measured by Heidelberg Spectralis, Zeiss Cirrus, or similar. | 6 months
  Evaluation of average RNFL thickness (µm).
Optical Coherence Tomography - Disc Rim Area, measured by Heidelberg Spectralis, Zeiss Cirrus, or similar. | 6 months
  Evaluation of Disc Rim Area (mm²).
Optical Coherence Tomography - Cup-to-disc Ratio, measured by Heidelberg Spectralis, Zeiss Cirrus, or similar. | 6 months
  Evaluation of Cup-to-disc ratio (average and vertical).
Optical Coherence Tomography - Central Subfield Thickness, measured by Heidelberg Spectralis, Zeiss Cirrus, or similar. | 6 months
  Evaluation of Central Subfield Thickness (µm).

SECONDARY OUTCOMES:
10 Visual Acuity, measured by Best Corrected Visual Acuity (BCVA) score, using Snellen and/or LogMar charts. | 6 months
  Changes in Best Corrected Visual Acuity (BCVA), Snellen and/or LogMar.
Adverse Events, as reported in patient's medical history. | 6 months
  Reported blurred vision, conjunctival hyperemia, dryness, itching, irritation, pain, light sensitivity, eye lash growth, changes in iris colour, orbital fat atrophy/periorbitopathy, intraocular inflammation, macular oedema, vitreous floaters.
Adherence to Study Treatment | 6 months
  Evaluation of number and percentage of participants adherence/compliance to study treatment (Yes or No).
Additional Glaucoma Interventions | 6 months
  Evaluation of number and percentage of occurrence of additional glaucoma-related procedures during the follow-up period [Laser trabeculoplasty and/or cataract surgery].

OTHER OUTCOMES:
Retinal Cells apoptosis Detected by DARC Imaging | 6 months
  Detection of Apoptosing Retinal Cells Cell Count
Vascular Outcomes - Change in the FAZ area (OCT-A parameter), measured by Zeiss Cirrus AngioPlex, or similar. | 6 months
  Detection and quantification of Apoptosing Retinal Cells Cell Count (e.g., cells/mm²)
Vascular outcomes - Change in Peripapillary Vessel Density (OCT-A parameter), measured by Zeiss Cirrus AngioPlex, or similar. | 6 months
  Evaluation of Peripapillary Vessel Density (%).
Vascular outcomes - Change in Macular Vessel Density (OCT-A parameter), measured by Zeiss Cirrus AngioPlex, or similar | 6 months
  Evaluation of Macular Vessel Density (mm-1).
Vascular outcomes - Change in perfusion density (OCT-A parameter), measured by Zeiss Cirrus AngioPlex, or similar. | 6 months
  Evaluation of perfusion density (a.u.).

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (2):
  - Department of Ophthalmology University of Bonn, Bonn
  - University Eye Hospital Leipzig, Leipzig
- Italy (2):
  - Centre for Clinical Trials at San Paolo Hospital University of Milan, Milan
  - Eye Unit, University Hospital Maggiore della Carità, Novara
- Spain (2):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Retina Unit, Department of Ophthalmology, Bellvitge University Hospital, Barcelona
- University Hospital Basel, Basel, Switzerland
- United Kingdom (3):
  - Clinical Eye Research Centre - St. Paul's Eye Unit, Royal Liverpool University Hospital, Liverpool
  - ICORG - Imperial College Ophthalmologic Research Group, London
  - NIHR Moorfields Clinical Research Facility, Moorfields Eye Hospital, NHS Foundation Trust, London

REFERENCES:
- [Background] Jonas JB, Aung T, Bourne RR, Bron AM, Ritch R, Panda-Jonas S. Glaucoma. Lancet. 2017 Nov 11;390(10108):2183-2193. doi: 10.1016/S0140-6736(17)31469-1. Epub 2017 May 31. PMID 28577860
- [Background] Leske MC, Heijl A, Hyman L, Bengtsson B, Dong L, Yang Z; EMGT Group. Predictors of long-term progression in the early manifest glaucoma trial. Ophthalmology. 2007 Nov;114(11):1965-72. doi: 10.1016/j.ophtha.2007.03.016. Epub 2007 Jul 12. PMID 17628686
- [Background] Peters D, Bengtsson B, Heijl A. Lifetime risk of blindness in open-angle glaucoma. Am J Ophthalmol. 2013 Oct;156(4):724-30. doi: 10.1016/j.ajo.2013.05.027. Epub 2013 Aug 7. PMID 23932216
- [Background] Chang EE, Goldberg JL. Glaucoma 2.0: neuroprotection, neuroregeneration, neuroenhancement. Ophthalmology. 2012 May;119(5):979-86. doi: 10.1016/j.ophtha.2011.11.003. Epub 2012 Feb 18. PMID 22349567
- [Background] Lee HP, Tsung TH, Tsai YC, Chen YH, Lu DW. Glaucoma: Current and New Therapeutic Approaches. Biomedicines. 2024 Sep 3;12(9):2000. doi: 10.3390/biomedicines12092000. PMID 39335514
- [Background] Yamamoto K, Sato K, Yukita M, Yasuda M, Omodaka K, Ryu M, Fujita K, Nishiguchi KM, Machida S, Nakazawa T. The neuroprotective effect of latanoprost acts via klotho-mediated suppression of calpain activation after optic nerve transection. J Neurochem. 2017 Feb;140(3):495-508. doi: 10.1111/jnc.13902. Epub 2016 Dec 27. PMID 27859240
- [Background] Yamagishi R, Aihara M, Araie M. Neuroprotective effects of prostaglandin analogues on retinal ganglion cell death independent of intraocular pressure reduction. Exp Eye Res. 2011 Sep;93(3):265-70. doi: 10.1016/j.exer.2011.06.022. Epub 2011 Jul 26. PMID 21791206
- [Background] Kanamori A, Naka M, Fukuda M, Nakamura M, Negi A. Latanoprost protects rat retinal ganglion cells from apoptosis in vitro and in vivo. Exp Eye Res. 2009 Mar;88(3):535-41. doi: 10.1016/j.exer.2008.11.012. Epub 2008 Dec 3. PMID 19084521
- [Background] Nakanishi Y, Nakamura M, Mukuno H, Kanamori A, Seigel GM, Negi A. Latanoprost rescues retinal neuro-glial cells from apoptosis by inhibiting caspase-3, which is mediated by p44/p42 mitogen-activated protein kinase. Exp Eye Res. 2006 Nov;83(5):1108-17. doi: 10.1016/j.exer.2006.05.018. Epub 2006 Jul 12. PMID 16839545
- [Background] Kudo H, Nakazawa T, Shimura M, Takahashi H, Fuse N, Kashiwagi K, Tamai M. Neuroprotective effect of latanoprost on rat retinal ganglion cells. Graefes Arch Clin Exp Ophthalmol. 2006 Aug;244(8):1003-9. doi: 10.1007/s00417-005-0215-0. Epub 2006 Jan 13. PMID 16411104
- [Background] Drago F, Valzelli S, Emmi I, Marino A, Scalia CC, Marino V. Latanoprost exerts neuroprotective activity in vitro and in vivo. Exp Eye Res. 2001 Apr;72(4):479-86. doi: 10.1006/exer.2000.0975. PMID 11273675
- [Background] Harper MM, Boese EA, Kardon RH, Ledolter J, Kuehn MH. High Correlation between Glaucoma Treatment with Topical Prostaglandin Analogs and BDNF Immunoreactivity in Human Retina. Curr Eye Res. 2021 May;46(5):739-745. doi: 10.1080/02713683.2020.1822417. Epub 2020 Sep 27. PMID 32985274
- [Background] Wagner IV, Stewart MW, Dorairaj SK. Updates on the Diagnosis and Management of Glaucoma. Mayo Clin Proc Innov Qual Outcomes. 2022 Nov 16;6(6):618-635. doi: 10.1016/j.mayocpiqo.2022.09.007. eCollection 2022 Dec. PMID 36405987
- [Background] Hill D, Choi S, Cordeiro MF. In Vivo Detection of Retinal Ganglion Cell Stress in Rodents with DARC. Methods Mol Biol. 2023;2708:123-129. doi: 10.1007/978-1-0716-3409-7_13. PMID 37558966
- [Background] Cordeiro MF, Hill D, Patel R, Corazza P, Maddison J, Younis S. Detecting retinal cell stress and apoptosis with DARC: Progression from lab to clinic. Prog Retin Eye Res. 2022 Jan;86:100976. doi: 10.1016/j.preteyeres.2021.100976. Epub 2021 Jun 5. PMID 34102318
- [Background] Yap TE, Donna P, Almonte MT, Cordeiro MF. Real-Time Imaging of Retinal Ganglion Cell Apoptosis. Cells. 2018 Jun 15;7(6):60. doi: 10.3390/cells7060060. PMID 29914056
- [Background] Stein JD, Khawaja AP, Weizer JS. Glaucoma in Adults-Screening, Diagnosis, and Management: A Review. JAMA. 2021 Jan 12;325(2):164-174. doi: 10.1001/jama.2020.21899. PMID 33433580
- [Background] Tan JC, Peters DM, Kaufman PL. Recent developments in understanding the pathophysiology of elevated intraocular pressure. Curr Opin Ophthalmol. 2006 Apr;17(2):168-74. doi: 10.1097/01.icu.0000193079.55240.18. PMID 16552252
- [Background] Conlon R, Saheb H, Ahmed II. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017 Feb;52(1):114-124. doi: 10.1016/j.jcjo.2016.07.013. Epub 2016 Nov 17. PMID 28237137
- [Background] Lee DA, Higginbotham EJ. Glaucoma and its treatment: a review. Am J Health Syst Pharm. 2005 Apr 1;62(7):691-9. doi: 10.1093/ajhp/62.7.691. PMID 15790795
- [Background] Toris CB, Gleason ML, Camras CB, Yablonski ME. Effects of brimonidine on aqueous humor dynamics in human eyes. Arch Ophthalmol. 1995 Dec;113(12):1514-7. doi: 10.1001/archopht.1995.01100120044006. PMID 7487618
- [Background] Toris CB, Gabelt BT, Kaufman PL. Update on the mechanism of action of topical prostaglandins for intraocular pressure reduction. Surv Ophthalmol. 2008 Nov;53 Suppl1(SUPPL1):S107-20. doi: 10.1016/j.survophthal.2008.08.010. PMID 19038618
- [Background] Chen JY, Le A, Caprioli J, Giaconi JA, Nouri-Mahdavi K, Law SK, Bonelli L, Coleman AL, Demer JL. Orbital Fat Volume After Treatment with Topical Prostaglandin Agonists. Invest Ophthalmol Vis Sci. 2020 May 11;61(5):46. doi: 10.1167/iovs.61.5.46. PMID 32455434
- [Background] Goh AS, Nassiri N, Kohn JC, Rootman DB, Giaconi J, Law SK, Coleman AL, Caprioli J, Goldberg RA. Prostaglandin Eyedrops Are Associated With Decreased Thicknesses of Eyelid Dermis and Orbicularis Oculi Muscle: Ultrasonographic Findings. Ophthalmic Plast Reconstr Surg. 2016 Sep-Oct;32(5):337-41. doi: 10.1097/IOP.0000000000000535. PMID 26237530
- [Background] Impagnatiello F, Bastia E, Almirante N, Brambilla S, Duquesroix B, Kothe AC, Bergamini MVW. Prostaglandin analogues and nitric oxide contribution in the treatment of ocular hypertension and glaucoma. Br J Pharmacol. 2019 Apr;176(8):1079-1089. doi: 10.1111/bph.14328. Epub 2018 May 24. PMID 29669171
- [Background] Sakata R, Shirato S, Miyata K, Aihara M. Incidence of deepening of the upper eyelid sulcus in prostaglandin-associated periorbitopathy with a latanoprost ophthalmic solution. Eye (Lond). 2014 Dec;28(12):1446-51. doi: 10.1038/eye.2014.224. Epub 2014 Sep 19. PMID 25233818
- [Background] Sakata R, Shirato S, Miyata K, Aihara M. Incidence of deepening of the upper eyelid sulcus on treatment with a tafluprost ophthalmic solution. Jpn J Ophthalmol. 2014 Mar;58(2):212-7. doi: 10.1007/s10384-013-0299-8. Epub 2014 Jan 7. PMID 24390604
- [Background] Fung TY, Iyaswamy A, Sreenivasmurthy SG, Krishnamoorthi S, Guan XJ, Zhu Z, Su CF, Liu J, Kan Y, Zhang Y, Wong HLX, Li M. Klotho an Autophagy Stimulator as a Potential Therapeutic Target for Alzheimer's Disease: A Review. Biomedicines. 2022 Mar 18;10(3):705. doi: 10.3390/biomedicines10030705. PMID 35327507
- [Background] Dong Q, Ding Y, Zhou Y, Zhao X, Hu L, Zhang Z, Xu X. Low-level expression of Cmyc in mature neurons: maintaining neuronal function and preventing neurodegeneration. Neural Regen Res. 2025 Apr 29. doi: 10.4103/NRR.NRR-D-24-01367. Online ahead of print. PMID 40313104
- [Background] Kang JM, Tanna AP. Glaucoma. Med Clin North Am. 2021 May;105(3):493-510. doi: 10.1016/j.mcna.2021.01.004. Epub 2021 Apr 2. PMID 33926643